CLINICAL TRIAL: NCT04377490
Title: Thrombo Embolic Events in Hospitalized Patients With Covid-19 Serious Acute Pneumopathy
Acronym: THROMBCOVID2
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2020_843_0040
Record Dates: First submitted 2020-05-05; First posted 2020-05-06 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: COVID-19; Hemostasis; Coagulation
Keywords: COVID-19; venous ultrasound; Hemostasis; coagulation
MeSH Terms: conditions — COVID-19; Thrombosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample for coagulation and hemostasis analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: venous ultrasound — Venous ultrasound will be performed on patients once a week, every week from the day of admission in Amiens Hospital until the day of patient discharge
Biological: blood sample — blood sample for coagulation and hemostasis analysis will be withdrawn from artery catheter from the day of admission in Amiens Hospital until the day of patient discharge

SUMMARY:
The understanding of haemostasis and inflammation cross-talk has gained considerable knowledge during the past decade in the field of arterial and venous thrombosis. Complex and delicately balanced interaction between coagulation and inflammation involve all cellular and humoral components.

Elements of the coagulation system such as activated thrombin, fibrinogen or factor Xa may increase inflammation by promoting the production of proinflammatory cytokines, chemokines, growth factors and adhesion molecules that lead to a procoagulant state amplifying the pathological process. Recent evidence supports inflammation as a common pathogenic contributor to both arterial and venous thrombosis, giving rise to the concept of inflammation induced thrombosis.

Patients with infection of COVID-19 and severe pneumoniae seem to have higher risk of thromboembolism. The purpose of this project is to analyze hemostasis and coagulation of every hospitalized patient with infection of COVID-19.

Blood sample for coagulation and hemostasis analysis will be collected on every patient hospitalized in Amiens hospital for COVID-19 infection. Thrombin time, factors V and II, fibrin/fibrinogen degradation products, antithrombin will be assessed every week. Anticardiolipin, anti-beta2 glycoprotein I and anti-annexin A2 antibodies IgG and IgM at day of admission and at fourth week after admission will be assessed. SARS-CoV2 viral load and serodiagnosis will be performed at the same time. At the same time venous ultrasound to diagnose thrombosis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* all patients hospitalized in Amiens Hospital with COVID-19 infection

Exclusion Criteria:

* patients< 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient hospitalized in CHU Amiens with COVID-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-05-04 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Variation of thrombin time (in secondes) in Hospitalized Covid-19 patients | up to 6 weeks
  Variation of thrombin time (in secondes) in Hospitalized Covid-19 patients. The reference range for the thrombin time is usually less than 20 seconds (ie, 15-19 seconds)
Variation of factor V concentration (U/dL) in Hospitalized Covid-19 patients. | up to 6 weeks
  Variation of factor V concentration (U/dL) in Hospitalized Covid-19 patients.
Variation of factor II concentration (U/dL) in Hospitalized Covid-19 patients | up to 6 weeks
  Variation of factor II concentration (U/dL) in Hospitalized Covid-19 patients
Variation of concentration of fibrin and fibrinogen degradation products (≥ 10 µgm/mL) in Hospitalized Covid-19 patients. | up to 6 weeks
  Variation of concentration of fibrin and fibrinogen degradation products (≥ 10 µgm/mL) in Hospitalized Covid-19 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Slama, Pr, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No